CLINICAL TRIAL: NCT00426543
Title: Phase 1 Study of B-cell Depletion With Rituximab on Oral, Ocular and General Disease Manifestations in Patients With Primary Sjögren's Syndrome
Brief Title: Effect of B-cell Depletion in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne Marie Lynge Pedersen, Associate Professor, PhD, DDS, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KF 02 282294; EudractCT-no. 2005-004740-31
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Primary Sjögren's Syndrome; Xerostomia; Hyposalivation; Keratoconjunctivitis Sicca; Fatigue
Keywords: Clinical trial; Intervention study; Double-blind randomised controlled study
MeSH Terms: conditions — Xerostomia; Keratoconjunctivitis Sicca; Fatigue | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MabThera (rituximab) — 1000 mg infusion twice with 14 days interval
  Other Names: Mabthera
Drug: Rituximab, Mabthera — 1000 mg Rituximab infusion in 500 ml isotonic sodiumchloride twice with 14 days interval

SUMMARY:
The primary purpose of the study is to determine whether B-cell depletion with Rituximab has an effect on the oral, ocular and general disease manifestations in patients with primary Sjögren´s syndrome, that is, an effect on the symptoms of oral and ocular dryness, improvement of the glandular function and a beneficial effect on the general symptoms such as fatigue. The secondary purpose of the study is the investigate the underlying autoimmune and pathophysiological mechanisms in Sjögren´s syndrome.

DETAILED DESCRIPTION:
The trial is designed as a double-blind parallel comparison between 2 infusions of 1 g Rituximab and solvent (saline) given two weeks apart, in 22 patients with the diagnosis of primary Sjögren's syndrome as based on the current American-European consensus classification criteria. The patients will be followed at the Department of Oral Medicine, Clinical Oral Physiology, Oral Pathology & Anatomy, University of Copenhagen, the Department of Rheumatology, Rigshospitalet and at the Department of Ophthalmology, Rigshospitalet.

The primary endpoints are clinical and a response has been delineated as at least 50% improvement in score. With the provision that this occurs for any item in at least 60% of the treated patients as compared to 1% in the control patients, a power of over 80% at doubled sided significance level of 5% is found with 20 patients.The patients will be followed within this study for 6 months after Rituximab.

The study will allow the first real dynamic appraisal of the immunologic pathophysiology in Sjögren's syndrome. Hence attempts will be made to determine at the best possible level if and how Rituximab influences and possibly resets the autoimmunity both at the whole body and particularly at the local level in the salivary glands. Also the basal transport mechanism in salivary secretion which must necessarily be perturbed in Sjögren's syndrome will be scrutinized employing the best available of techniques. Every possible effort to envisage a priory, and then monitor, the decisive mechanisms has been made.

In particular this includes repetitive biopsies from the parotid glands, which will allow combining functional and structural data to reduce as much as possible random variability of crucial quantities. Also this will allow for the first time to assess the relative and combined utility of obtaining biopsies from both the parotid and labial salivary glands.

Roche A/S provide investigational medicine, but the study was initiated and is entirely controlled by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Female patients fulfilling the current American-European consensus classification criteria.
* Fertile-age female patients must use safe anticonceptional methods such as pills, mini-pills, or intrauterine spiral.
* The fertile-age females included in the study must not get pregnant in at least 12 months after the last treatment with Rituximab.

Exclusion Criteria:

* Pregnancy and lactation.
* Fertile-age females who do not use safe anticonceptional methods.
* Patients in systemic treatment with cytostatics.
* Patients who previously have been treated with Rituximab.
* Patient with an active infection that requires antibiotic treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of Rituximab on subjective disease symptoms including oral dryness, ocular dryness, myoartralgia and fatigue. | Baseline, Day 22 after second treatment, 1 month, 3 months and 6 months after treatment.

SECONDARY OUTCOMES:
To study the effect of Rituximab: on the structural changes (focal lymphocytic infiltrates) in the labial salivary gland tissue, including changes in the T- and B-cell ratio in the infiltrates as well as in the expression of M3-receptors | Baseline and 6 months after treatment
On the salivary gland function, incl. the production and composition of whole saliva and parotid saliva, the cellular signalling mechanisms and also the distribution of M3-receptors (M3R), the expression of aquaporins, | Baseline, 1 month, 3 months and 6 months after treatment
On the circulating serum autoantibodies (anti-SSA/-SSB, rheumatoid factors) and on antibodies against the M3R and α-fodrin and on the IgG level. | Baseline, 1 month, 3 months and 6 months after treatment
On the phenotype of circulating T- and B-cells as well as cytokines and immunoregulators, especially BLyS/BAFF. | Baseline, 1 month, 3 months and 6 months after treatment
On the function of the tear glandula, including the quantity and quality of tear as well as the extent of corneal changes. | Baseline, 1 month, 3 months and 6 months after treatment
To evaluate the side-effects in relation to the use of Rituximab-/placebo treatment. | After first and second treatment and after 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Lynge Pedersen, PhD, DDS, Principal Investigator — Institute of Odontology, Faculty of Health Sciences, University of Copenhagen
Locations (1):
- Institute of Odontology, Faculty of Health Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Ring T, Kallenbach M, Praetorius J, Nielsen S, Melgaard B. Successful treatment of a patient with primary Sjogren's syndrome with Rituximab. Clin Rheumatol. 2006 Nov;25(6):891-4. doi: 10.1007/s10067-005-0086-0. Epub 2005 Nov 8. PMID 16283417